CLINICAL TRIAL: NCT03980145
Title: G-EO Gait Rehabilitation Training in Progressive Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: University of Alabama at Birmingham (Other); University of Ottawa (Other)
Responsible Party: Principal Investigator, Peter Altenburger, Associate Professor, Health and Rehabilitation, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1701909134
Record Dates: First submitted 2019-02-26; First posted 2019-06-10 (Actual); Results first posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Progressive Multiple Sclerosis
Keywords: Robotics; Gait Training
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Conventional Physical Therapy (Active Comparator): Conventional physical therapy (CPT): CPT sessions will involve a 3-5 minute warm-up, stretching, progressive strength training exercises, and gait and balance training.40-43 Additional strategies for home exercises, energy conservation, fall prevention, and appropriate assistive devices (i.e., orthotics) will be provided.
  Interventions: Other: Conventional Physical Therapy
- End-Effector Robotic Training (Experimental): G-EO training: Using the G-EO System, participants will be secured with the appropriate sized harness and attached to an overhead body-weight support system, with feet secured to pressure sensitive footplates. Each session will begin with a 3-5 minute warm-up in the continuous passive mode (cadence ~40-45 steps/minute). The participant will then be transitioned into the adaptive training phase for practicing repetitive floor walking and stair climbing for up to 30 minutes. During this phase, the force produced by the robot is modulated to support the effort of the patient in producing a typical walking pattern.
  Interventions: Device: G-EO System (Reha Technology AG: Olten, Switzerland)

INTERVENTIONS:
Device: G-EO System (Reha Technology AG: Olten, Switzerland) — Electromechanically-assisted gait training addresses many of the limitations of therapist-assisted gait training and can be performed using either exoskeleton or end-effector devices. Exoskeleton devices involve programmable drives or passive elements which physically move the lower limbs, whereas, end-effector approaches involve driven footplates that have trajectories that simulate the stance and swing phases.13,14 The G-EO System (Reha Technology: Olten, Switzerland) is a novel end-effector gait training system that was developed for regaining mobility and independence in stroke survivors. This system involves minimal therapist and patient burden (e.g., quick set-up, single operate usage), there is the unique capacity for practicing walking and stair climbing movements, and the patient can receive real-time visual feedback.
  Other Names: Electromechanically-assisted gait training; Robotic end-effector gait training system
  Arms: End-Effector Robotic Training
Other: Conventional Physical Therapy — Conventional physical therapy (CPT): CPT sessions will involve a 3-5 minute warm-up, stretching, progressive strength training exercises, and gait and balance training. Additional strategies for home exercises, energy conservation, fall prevention, and appropriate assistive devices (i.e., orthotics) will be provided.
  Arms: Conventional Physical Therapy

SUMMARY:
The logistic advantages and advanced training capabilities of the G-EO System, as well as the benefits reported in other populations, support this strategy as a potentially potent rehabilitation tool for restoring and maintaining function in progressive Multiple Sclerosis (MS). This approach represents a paradigm shifting opportunity for improving current clinical practices for patients with progressive MS. If successful, this project will provide initial evidence for increasing patient access to the G-EO System, and this could be accomplished through "regional technology centers" using a rural health-delivery approach.

There are several novel aspects of the proposed trial: (1) the examination of a novel gait rehabilitation stimulus (G-EO System) that could alter current clinical practices; (2) the focus on patients with progressive MS who have gait impairment (i.e., those who have received minimal research attention), which was recently described as the greatest therapeutic challenge facing the MS community; and (3) a study design that accounts for standard therapy.

Specific Aims: The investigators designed a single-blinded, randomized pilot trial of electromechanically-assisted gait training using the G-EO System in patients with progressive MS with gait disability (EDSS=4.0-7.5).

Specific Aim 1 will establish the safety and feasibility of gait training using the G-EO System.

Specific Aim 2 will determine the efficacy of gait training using the G-EO System for improving mobility, symptomatic, quality of life, and participatory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years
* Confirmed diagnosis of Primary or Secondary Progressive Multiple Sclerosis (this will be confirmed by the referring physician)
* EDSS 4.0-7.522
* Stable course of disease-modifying therapy over the past 6 months
* Asymptomatic (i.e., no underlying cardiovascular disease)
* Physician approval for exercise
* Willingness to visit the IU Health Neurosciences Center for testing and training

Exclusion Criteria:

* Pregnancy
* Current use of dalfampridine (Ampyra®)
* Conventional physical therapy or G-EO training within the past 6 months
* Height <1m or >2m
* Body weight >150 kg
* Contraindications to G-EO gait training (e.g., bone instability)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Altenburger, PhD, PT, Principal Investigator — Indiana University
Locations (1):
- Neurorehabilitation and Robotics at IU Health Neuroscience Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- End-Effector Robotic Training: G-EO training: Using the G-EO System, participants will be secured with the appropriate sized harness and attached to an overhead body-weight support system, with feet secured to pressure sensitive footplates. Each session will begin with a 3-5 minute warm-up in the continuous passive mode (cadence ~40-45 steps/minute). The participant will then be transitioned into the adaptive training phase for practicing repetitive floor walking and stair climbing for up to 30 minutes. During this phase, the force produced by the robot is modulated to support the effort of the patient in producing a typical walking pattern.
  G-EO System (Reha Technology AG: Olten, Switzerland): Electromechanically-assisted gait training addresses many of the limitations of therapist-assisted gait training and can be performed using either exoskeleton or end-effector devices. Exoskeleton devices involve programmable drives or passive elements which physically move the lower limbs, whereas, end-effector approaches involve driven footplates that have trajectories that simulate the stance and swing phases.13,14 The G-EO System (Reha Technology: Olten, Switzerland) is a novel end-effector gait training system that was developed for regaining mobility and independence. This system has a unique capacity for practicing walking and stair climbing movements, and the patient can receive real-time visual feedback.
Period: Overall Study
Arm/Group | Conventional Physical Therapy | End-Effector Robotic Training
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- End-Effector Robotic Training: G-EO training: Using the G-EO System, participants will be secured with the appropriate sized harness and attached to an overhead body-weight support system, with feet secured to pressure sensitive footplates. Each session will begin with a 3-5 minute warm-up in the continuous passive mode (cadence ~40-45 steps/minute). The participant will then be transitioned into the adaptive training phase for practicing repetitive floor walking and stair climbing for up to 30 minutes. During this phase, the force produced by the robot is modulated to support the effort of the patient in producing a typical walking pattern.
  G-EO System (Reha Technology AG: Olten, Switzerland): Electromechanically-assisted gait training addresses many of the limitations of therapist-assisted gait training and can be performed using either exoskeleton or end-effector devices. Exoskeleton devices involve programmable drives or passive elements which physically move the lower limbs, whereas, end-effector approaches involve driven footplates that have trajectories that simulate the stance and swing phases. The G-EO System (Reha Technology: Olten, Switzerland) is a novel end-effector gait training system that was developed for regaining mobility and independence. This system has the capacity for practicing walking and stair climbing movements, and the patient can receive real-time visual feedback.
- Total: Total of all reporting groups
Arm/Group | Conventional Physical Therapy | End-Effector Robotic Training | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (11.58) | 49.4 (14.46) | 52.5 (13.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 3 | 1 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15
Expanded Disability Status Scale (EDSS) [Mean (Standard Deviation); unit: units on a scale] — The Expanded Disability Status Scale is used to quantify disability in individuals with Multiple Sclerosis The scale ranges from 0 to 10 and is used to monitor an individuals changing level of disability throughout their lifetime. A higher score represents greater disability. Scores ranging between 1 and 5 indicated minimal or no impact on walking while scores greater than 5 have progressively more impact on walking ability.
  units on a scale | 6.0 (0.33) | 5.81 (0.88) | 5.9 (0.74)

OUTCOME MEASURES:

1. Primary Outcome: Comfortable Walking Speed
Description: Comfortable Walking speed will be assessed using a Pressure Sensor Walkway. Participants will be asked to walk over a 14 foot pressure mat that will capture their walking speed. Scores range from 0 (no speed) to as fast as they are comfortable with the most common range being .1 to 1.5 meters per second.
Time Frame: Gait speed for comfortable walking will be assessed prior to the start of the treatment (Pretest) and following study completion which occurred following 20 treatment visits (Posttest)
Measure: Mean (Standard Error); unit: meters per second
Arm/Group | Conventional Physical Therapy | End-Effector Robotic Training
Number analyzed (Participants) | 7 | 8
meters per second
  Pretest Assessment (Prior to starting intervention training) | .45 (.080) | .60 (.137)
  Posttest Assessment (After completing intervention training) | .52 (0.90) | .67 (.163)
Statistical Analysis 1: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Null hypothesis is no difference between the two groups; Test type: Superiority; p = .405, ANOVA — Statistical significance set at .05
Statistical Analysis 2: Comparison: End-Effector Robotic Training; Null hypothesis is no difference between pretest and posttest; Test type: Superiority; p = .133, ANOVA
Statistical Analysis 3: Comparison: Conventional Physical Therapy; Evaluated the difference between the pretest and posttest within the conventional physical therapy group; Test type: Superiority; p = .050, ANOVA
Statistical Analysis 4: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Evaluating the impact of whether comfortable walking speed for both groups combined resulted in a significant improvement in walking speed; Test type: Superiority; p = .017, ANOVA — p value was adjusted for multiple comparisons using a Bonferroni correction; Mean Difference (Final Values) = .070, 95% CI 2-sided [.015 to .124]

2. Primary Outcome: Two Minute Walk Test
Description: A 2-minute walk (2MWT) test to determine walking endurance. Subjects will be asked to walk for 2 minutes along a 30m track. Subjects may stop and rest as often as needed. The outcome is the distance in meters traveled during the 2 minutes. Scores can range from 0 to 500 meters. An increase in distance following treatment when compared to pretest numbers would indicate improved muscular and cardiovascular endurance.
Time Frame: Walking distance will be assessed prior to the start of the treatment (Pretest) and following study completion (Posttest). Pretest represents a time point prior to intervention training. Posttest represents the point following intervention completion.
Measure: Mean (Standard Error); unit: Meters
Groups:
- End-Effector Robotic Training: G-EO training: Using the G-EO System, participants will be secured with the appropriate sized harness and attached to an overhead body-weight support system, with feet secured to pressure sensitive footplates. Each session will begin with a 3-5 minute warm-up in the continuous passive mode (cadence ~40-45 steps/minute). The participant will then be transitioned into the adaptive training phase for practicing repetitive floor walking and stair climbing for up to 30 minutes.
  G-EO System (Reha Technology AG: Olten, Switzerland): Electromechanically-assisted gait training addresses many of the limitations of therapist-assisted gait training and can be performed using either exoskeleton or end-effector devices. Exoskeleton devices involve programmable drives or passive elements which physically move the lower limbs, whereas, end-effector approaches involve driven footplates that have trajectories that simulate the stance and swing phases. The G-EO System (Reha Technology: Olten, Switzerland) is a novel end-effector gait training system that was developed for regaining mobility and independence. This system has the capacity for practicing walking and stair climbing movements, and the patient can receive real-time visual feedback.
Arm/Group | Conventional Physical Therapy | End-Effector Robotic Training
Number analyzed (Participants) | 7 | 8
Meters
  Pretest Assessment (Prior to the start of intervention training) | 66.57 (10.90) | 89.35 (21.38)
  Posttest Assessment (Following completion of intervention training) | 72.62 (14.23) | 93.21 (19.14)
Statistical Analysis 1: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Comparison of the impact between the two arms looking an improved walking endurance; Test type: Superiority; p = .369, ANOVA
Statistical Analysis 2: Comparison: End-Effector Robotic Training; Evaluation of impact of end-effector robotic training alone; Test type: Superiority; p = .710, ANOVA
Statistical Analysis 3: Comparison: Conventional Physical Therapy; Evaluating the impact of conventional therapy on walking endurance Null hypothesis is no difference between pretest and posttest; Test type: Superiority; p = .682, ANOVA
Statistical Analysis 4: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Evaluating the impact of whether both groups combined resulted in a significant change in walking distance; Test type: Superiority; p = .568, ANOVA — p value adjusted for multiple comparisons - Bonferroni

3. Primary Outcome: Modified Fatigue Impact Scale
Description: Subjects will complete a questionnaire evaluating their level of perceived fatigue. The scores are divided into three different scales: physical, cognitive, and psychosocial. A total score is also calculated. Scale scores are represented by the following ranges: physical subscale ranges from 0 to 36; cognitive subscale from 0 to 40; and psychosocial subscale from 0 to 8. A total score has a range of 0 to 85. A higher score indicates greater fatigue. Decreases in scores over time indicate decreases in feelings of fatigue. Each scale including the total score is summed.
Time Frame: Subjects perception of the their fatigue will be assessed prior to the start of the treatment and following study completion (at 10 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- End-Effector Robotic Training: G-EO training: Using the G-EO System, participants will be secured with the appropriate sized harness and attached to an overhead body-weight support system, with feet secured to pressure sensitive footplates. Each session will begin with a 3-5 minute warm-up in the continuous passive mode (cadence ~40-45 steps/minute). The participant will then be transitioned into the adaptive training phase for practicing repetitive floor walking and stair climbing for up to 30 minutes.
  G-EO System (Reha Technology AG: Olten, Switzerland): Electromechanically-assisted gait training addresses many of the limitations of therapist-assisted gait training and can be performed using either exoskeleton or end-effector devices. Exoskeleton devices involve programmable drives or passive elements which physically move the lower limbs, whereas, end-effector approaches involve driven footplates that have trajectories that simulate the stance and swing phases.13,14 The G-EO System (Reha Technology: Olten, Switzerland) is a novel end-effector gait training system that was developed for regaining mobility and independence in stroke survivors. This system involves minimal therapist and patient burden (e.g., quick set-up, single operate usage), there is the unique capacity for practicing walking and stair climbing movements, and the patient can receive real-time visual feedback.
Arm/Group | Conventional Physical Therapy | End-Effector Robotic Training
Number analyzed (Participants) | 7 | 8
score on a scale
  Pretest Total Score | 50.14 (4.93) | 43.75 (4.61)
  Posttest Total Score | 40.71 (5.20) | 34.25 (4.87)
  Pretest Physical Domain | 23.71 (3.74) | 25.88 (1.74)
  Posttest Physical Domain | 24.57 (1.55) | 19.50 (2.33)
  Pretest Cognitive Domain | 20.43 (1.78) | 14.37 (4.04)
  Posttest Cognitive Domain | 12.14 (2.86) | 11.88 (3.54)
  Pretest Psychological Domain | 6.0 (.436) | 3.50 (.964)
  Posttest Psychological Domain | 4.0 (.535) | 2.88 (.766)
Statistical Analysis 1: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Evaluation of the physical domain; Test type: Superiority; p = .594, ANOVA — Outcome specific to the physical domain
Statistical Analysis 2: Comparison: End-Effector Robotic Training; Pretest- Posttest End Effector Robotic Training Comparison for the Physical Domain; Test type: Superiority; p = .061, ANOVA
Statistical Analysis 3: Comparison: Conventional Physical Therapy; Pretest posttest comparison of conventional training group for physical domain; Test type: Superiority; p = .812, ANOVA
Statistical Analysis 4: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Combined conventional and end-effector training for outcomes in the physical domain; Test type: Superiority; p = .235, ANOVA
Statistical Analysis 5: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Between group assessment of changes in the MFIS Cognitive domain; Test type: Superiority; p = .465, ANOVA
Statistical Analysis 6: Comparison: End-Effector Robotic Training; Within group differences for the End Effector Robotic Training Group for the Cognitive Domain; Test type: Superiority; p = .165, ANOVA
Statistical Analysis 7: Comparison: Conventional Physical Therapy; Within group assessment for the conventional group within the cognitive domain of the MFIS; Test type: Superiority; p = .682, ANOVA
Statistical Analysis 8: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Combined group outcomes comparing pretest to posttest for the cognitive domain; Test type: Superiority; p = .017, ANOVA — p value adjusted using a Bonferroni correction; Mean Difference (Final Values) = 5.39, 95% CI 2-sided [1.12 to 9.67]
Statistical Analysis 9: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Between group comparison for the MFIS Psychological Subscale; Test type: Superiority; p = .052, ANOVA
Statistical Analysis 10: Comparison: End-Effector Robotic Training; Within group comparison for the end-effector robotic training group for the MFIS Psychological subscale; Test type: Superiority; p = .483, ANOVA
Statistical Analysis 11: Comparison: Conventional Physical Therapy; Within group assessment for the conventional physical therapy group for the MFIS Psychological subscale; Test type: Superiority; p = .056, ANOVA
Statistical Analysis 12: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Change in MFIS for all subjects from pre to posttest for the psychological subscale; Test type: Superiority; p = .048, ANOVA — p value is adjusted for multiple comparisons using a Bonferroni correction; Mean Difference (Final Values) = 1.313, 95% CI 2-sided [.016 to 2.619]
Statistical Analysis 13: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Between group assessment of differences in total score; Test type: Superiority; p = .010, ANOVA
Statistical Analysis 14: Comparison: End-Effector Robotic Training; Within assessment of change in total fatigue score; Test type: Superiority; p = .089, ANOVA
Statistical Analysis 15: Comparison: Conventional Physical Therapy; Within group assessment of change in total score; Test type: Superiority; p = .50, ANOVA
Statistical Analysis 16: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Combined assessment of all subject improvement in total MFIS score; Test type: Superiority; p = 0.10, ANOVA; Mean Difference (Final Values) = 9.464, 95% CI 2-sided [2.678 to 16.251]

4. Primary Outcome: Multiple Sclerosis Impact Scale-29
Description: Subjects completed a 29 item questionnaire evaluating their level of health-related quality of life. The higher the score the greater the impact MS is having on their daily function. The 29 items are divided into a 20 item physical scale and 9 item psychological scale. Each item has four potential responses resulting in scores on the physical impact scale ranging from 20 to 80 and on the psychological impact scale ranging from 9 to 36. Final scores for each scale are achieved by summing the items for each of the two scales and then transforming them to a 100 point scale for easy comparison. On the 100 point scale, 0 would indicate no impact of the disease on daily function and 100 would indicate the greatest possible impact.
Time Frame: Subjects perception of the their disability will be assessed prior to the start of the treatment and following study completion (at 10 weeks)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Conventional Physical Therapy | End-Effector Robotic Training
Number analyzed (Participants) | 7 | 8
units on a scale
  Pretest Physical Subscale | 65.89 (4.26) | 47.97 (7.97)
  Posttest Physical Subscale | 52.32 (5.14) | 33.13 (8.14)
  Pretest Psychological Subscale | 55.16 (3.12) | 30.56 (7.57)
  Posttest Psychological Subscale | 32.94 (3.34) | 26.39 (7.84)
Statistical Analysis 1: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Null hypothesis set for no difference between groups Assessment of between group differences for the physical subscale; Test type: Superiority; p = .071, ANOVA
Statistical Analysis 2: Comparison: End-Effector Robotic Training; With group assessment of change on the physical subscale of the MSIS; Test type: Superiority; p = .005, ANOVA; Mean Difference (Final Values) = 14.84, 95% CI 2-sided [6.02 to 23.66]
Statistical Analysis 3: Comparison: Conventional Physical Therapy; With group assessment of change on the physical subscale of the MSIS; Test type: Superiority; p = .001, ANOVA; Mean Difference (Final Values) = 13.57, 95% CI 2-sided [8.30 to 18.85]
Statistical Analysis 4: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Combined group assessment of change on the physical subscale of the MSIS; Test type: Superiority; p = .000026, ANOVA — p value adjusted for multiple comparisons using Bonferroni; Mean Difference (Final Values) = 14.21, 95% CI 2-sided [9.367 to 19.04]
Statistical Analysis 5: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Between group comparison for the psychological subscale for the MSIS; Test type: Superiority; p = .084, ANOVA — Pretest measures were statistically different between the two groups
Statistical Analysis 6: Comparison: End-Effector Robotic Training; Within group comparison for the psychological subscale for the MSIS; Test type: Superiority; p = .412, ANOVA
Statistical Analysis 7: Comparison: Conventional Physical Therapy; Within group comparison for the psychological subscale for the MSIS; Test type: Superiority; p = .00018, ANOVA; Mean Difference (Final Values) = 22.22, 95% CI 2-sided [15.59 to 28.85]
Statistical Analysis 8: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Combined group comparison for the psychological subscale for the MSIS; Test type: Superiority; p = .00049, ANOVA; Mean Difference (Final Values) = 13.19, 95% CI 2-sided [7.013 to 19.38]

5. Primary Outcome: Fast Walking Speed
Description: Fast Walking speed will be assessed using a Pressure Sensor Walkway. Participants will be asked to walk over a 14 foot pressure mat that will capture their walking speed. Scores range from 0 (no speed) to as fast as they are able with the most common range being .5 to 2.0 meters per second.
Time Frame: Fast walking speed will be assessed prior to the start of the treatment (Pretest) and following study completion (Posttest). Pretest represents a time point prior to intervention training. Posttest represents the point following intervention completion.
Measure: Mean (Standard Error); unit: meters per second
Arm/Group | Conventional Physical Therapy | End-Effector Robotic Training
Number analyzed (Participants) | 7 | 8
meters per second
  Pretest Assessment (Prior to intervention training) | .55 (.108) | .81 (.190)
  Posttest Assessment (following completion of intervention training) | .63 (.131) | .84 (.205)
Statistical Analysis 1: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Null hypothesis is no difference between the two groups; Test type: Superiority; p = .352, ANOVA
Statistical Analysis 2: Comparison: Conventional Physical Therapy; Within group assessment; Test type: Superiority; p = .079, ANOVA
Statistical Analysis 3: Comparison: End-Effector Robotic Training; Within group assessment; Test type: Superiority; p = .393, ANOVA
Statistical Analysis 4: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Evaluating the impact of whether fast walking speed for both groups combined resulted in a significant improvement in walking speed; Test type: Superiority; p = .048, ANOVA; Adjusted for multiple mean comparisons; Mean Difference (Final Values) = .058, 95% CI 2-sided [.001 to .116]

6. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: Subjects completed a questionnaire evaluating their level of anxiety and depression. The questionnaire is comprised of two scales: a 7 item scale related to anxiety and 7 item scale related to depression. Each item within both scales is scored using a 0-3 scoring system depending upon the individual's answer. Both the anxiety scale and the depression scale can range in scores from 0 to 21. Although the 14 items were administered together, each set of seven questions was kept separate and scored separately to create a score for anxiety and one for depression. The scores for each scale were summed to provide a total score for anxiety and a separate score for depression. The higher the score the greater the severity. A score between 8-10 is consider mild, 11-14 is moderate, >14 is severe for both scales.
Time Frame: Subjects perception of the their anxiety and depression will be assessed prior to the start of the treatment and following study completion (at 10 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Conventional Physical Therapy | End-Effector Robotic Training
Number analyzed (Participants) | 7 | 8
score on a scale
  Pretest HADS Anxiety Score | 8.43 (1.445) | 5.88 (1.076)
  Posttest HADS Anxiety Score | 7.14 (1.223) | 4.75 (1.161)
  Pretest HADS Depression Score | 7.57 (.869) | 4.75 (1.187)
  Posttest HADS Depression Score | 7.00 (.845) | 3.88 (1.445)
Statistical Analysis 1: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Between group assessment for the HADS Anxiety Subscale; Test type: Superiority; p = .117, ANOVA
Statistical Analysis 2: Comparison: End-Effector Robotic Training; Within group assessment for HADS Anxiety Subscale; Test type: Superiority; p = .041, ANOVA; Mean Difference (Final Values) = 1.75, 95% CI 2-sided [.093 to 3.407]
Statistical Analysis 3: Comparison: Conventional Physical Therapy; Within group assessment for HADS Anxiety Subscale; Test type: Superiority; p = .150, ANOVA
Statistical Analysis 4: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Combined group assessment of HADS Anxiety Subscale; Test type: Superiority; p = .012, ANOVA — p value adjusted for multiple comparisons; Mean Difference (Final Values) = 1.518, 95% CI 2-sided [.390 to 2.646]

7. Secondary Outcome: Short Form McGill Pain Questionnaire
Description: Subjects completed a questionnaire evaluating their level of pain. There are 15 adjectives that describe the patient's pain. The patient ranks each of the words on a categoric scale of "none, mild, moderate, severe. Sensory and affective scores will be computed separately. Scores are created from a summary of the responses using an intensity scale of 0 = none, 1 = mild, 2 = moderate and 3 = severe. The higher the score the more severe the pain is for each of the subscales. For this study, sensory, affective, and total pain scores are reported. The minimum sensory, affective, and total score score would be zero. The maximum score for sensory is 33, affective is 12, and total is 45.
Time Frame: Subjects perception of the their pain will be assessed prior to the start of the treatment and following study completion (at 10 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Conventional Physical Therapy | End-Effector Robotic Training
Number analyzed (Participants) | 7 | 8
score on a scale
  Pretest Sensory Pain | 10.14 (2.80) | 5.00 (2.62)
  Posttest Sensory Pain | 8.29 (2.88) | 5.38 (2.70)
  Pretest Affective Pain | 2.57 (.80) | 1.63 (.74)
  Posttest Affective Pain | 2.29 (1.22) | 1.88 (1.15)
  Pretest Total Pain | 12.71 (4.057) | 6.63 (2.890)
  Posttest Total Pain | 11.14 (4.114) | 7.25 (4.057)
Statistical Analysis 1: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Test type: Superiority; p = .239, ANOVA
Statistical Analysis 2: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Comparison between groups for differences in sensory pain score; Test type: Superiority; p = .667, ANOVA
Statistical Analysis 3: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Between group differences in affective pain; Test type: Superiority; p = .770, ANOVA

8. Secondary Outcome: Late-Life Disability Inventory (LLFDI)
Description: Subjects will complete a questionnaire evaluating their perceived level of disability. This tool assesses and responds to meaningful change in a persons disability (Ability to participate in life's activities). There is a 16 item disability component that is scored across two dimensions: frequency and limitation. Total scores and dimensional scores are created by summation and conversion to a 100 point scaled score. The instrument provides a table for converting the raw score to a scaled score. The lowest possible scale score is 0 and the highest score is 100 for both frequency and limitation. A higher score indicates greater functional ability and less disability.
  Each dimension can be further assessed by analyzing domains. There are social and personal domains within the frequency dimension and instrumental and management domains within the limitations dimension. All domains are calculated as described before through summation and scale adjustment.
Time Frame: Subjects perception of the their functional ability using the total score and dimensional scores will be assessed prior to the start of the treatment and following study completion (at 10 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Conventional Physical Therapy | End-Effector Robotic Training
Number analyzed (Participants) | 7 | 8
score on a scale
  LLFDI Frequency Pretest | 50.10 (2.13) | 55.21 (2.38)
  LLFDI Frequency Posttest | 49.78 (2.74) | 54.93 (2.57)
  LLFDI Limitations Pretest | 52.72 (1.79) | 60.27 (2.73)
  LLFDI Limitations Posttest | 56.00 (2.78) | 62.44 (2.99)
Statistical Analysis 1: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Between group assessment of LLFDI Disability Frequency; Test type: Superiority; p = .136, ANOVA
Statistical Analysis 2: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Combined group assessment of improvement in LLFDI Disability Frequency; Test type: Superiority; p = .833, ANOVA
Statistical Analysis 3: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Between Group Assessment of improvement in LLFDI Disability Limitations; Test type: Superiority; p = .044, ANOVA; Mean Difference (Final Values) = 6.996, 95% CI 2-sided [.212 to 13.781]
Statistical Analysis 4: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Combined group assessment of improvement in LLFDI Disability Limitations; Test type: Superiority; p = .212, ANOVA

9. Secondary Outcome: Late-Life Function Inventory
Description: Subjects will complete a questionnaire evaluating their perceived level of function. This tool assesses and responds to meaningful change in a persons function (ability to execute discrete tasks). There is a 32 item functional component is comprised of three domains Upper Extremity, Basic Lower Extremity, Advanced Lower Extremity. Total score and each domain will be scored by summing and then converting to a 100 point scaled score. The instrument provides a table for converting the raw score to a scaled score. A higher score indicates greater functional ability. The lowest score would be 0 and the highest scale score would be 100.
Time Frame: Subjects perception of the their functional ability using all three domains will be assessed prior to the start of the treatment and following study completion (at 10 weeks)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Conventional Physical Therapy | End-Effector Robotic Training
Number analyzed (Participants) | 7 | 8
score on a scale
  LLDFI Function Pretest | 43.65 (1.51) | 45.76 (2.96)
  LLFDI Function Posttest | 48.13 (2.70) | 53.27 (3.24)
Statistical Analysis 1: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Between group comparison for the LLDFI Function; Test type: Superiority; p = .338, ANOVA
Statistical Analysis 2: Comparison: End-Effector Robotic Training; Within group assessment of LLFDI Function; Test type: Superiority; p = .007, ANOVA; Mean Difference (Final Values) = 7.508, 95% CI 2-sided [2.73 to 12.28]
Statistical Analysis 3: Comparison: Conventional Physical Therapy; Within group assessment for changes in LLFDI Function; Test type: Superiority; p = .067, ANOVA
Statistical Analysis 4: Comparison: Conventional Physical Therapy vs End-Effector Robotic Training; Combined group improvement in LLFDI Function; Test type: Superiority; p = .001, ANOVA — p value adjusted for multiple comparisons; Mean Difference (Final Values) = 5.99, 95% CI 2-sided [2.90 to 9.08]

ADVERSE EVENTS:
Time Frame: 10 weeks
Groups:
- End-Effector Robotic Training: G-EO training: Using the G-EO System, participants will be secured with the appropriate sized harness and attached to an overhead body-weight support system, with feet secured to pressure sensitive footplates. Each session will begin with a 3-5 minute warm-up in the continuous passive mode (cadence ~40-45 steps/minute).
  G-EO System (Reha Technology AG: Olten, Switzerland): Electromechanically-assisted gait training addresses many of the limitations of therapist-assisted gait training and can be performed using either exoskeleton or end-effector devices. Exoskeleton devices involve programmable drives or passive elements which physically move the lower limbs, whereas, end-effector approaches involve driven footplates that have trajectories that simulate the stance and swing phases. The G-EO System (Reha Technology: Olten, Switzerland) is a novel end-effector gait training system that was developed for regaining mobility and independence. This system has the capacity for practicing walking and stair climbing movements, and the patient can receive real-time visual feedback.
Arm/Group | Conventional Physical Therapy | End-Effector Robotic Training
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT03980145/Prot_SAP_000.pdf